CLINICAL TRIAL: NCT03648918
Title: Genetics Of Autoimmunity In Type I Diabetes
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Benaroya Research Institute (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Martin Hessner, Professor, Medical College of Wisconsin
Other Study IDs: 142618; McGee Sibling Study (Other: Medical College of Wisconsin)
Record Dates: First submitted 2018-04-16; First posted 2018-08-28 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Type1diabetes; Diabetes Mellitus, Type 1; Type1 Diabetes Mellitus; Diabetes Mellitus
Keywords: Family; Healthy Controls; Siblings
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The investigators will be collecting blood samples, which will be analyzed for HLA haplotype (a genetic sequence related to type 1 diabetes susceptibility), plasma-induced signature, diabetes autoantibodies, and complete blood count with differential, as well as plasma for storage. Blood will be analyzed for A1c for participants with diabetes. Specimens will be used and stored until none is left.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Blood Collection — Blood will be collected via venipuncture and analyzed. Blood samples will be analyzed for HLA haplotype (a genetic sequence related to type 1 diabetes susceptibility), plasma-induced signature, diabetes autoantibodies, complete blood count with differential, and serum and plasma for storage. For family members with diabetes, blood will also be tested for A1c.

SUMMARY:
The purpose of this study is to gain more information about the step-by-step process that causes someone to develop type 1 diabetes. Scientists think that a person's own immune system, directed by genetic and environmental factors play a major role in its development. Participation involves a blood draw, a brief medical history questionnaire and measurements of height and weight. Some participants will be asked to return for annual follow-up visits for 10 years.

DETAILED DESCRIPTION:
The goal of this project is to gain knowledge about the development of Type 1 diabetes (T1D), as T1D is one of the most common chronic diseases in children. There has been a rise in the number of cases diagnosed as well as a decrease in the age of diagnosis. This project aims to understand the disease progression as seen in the immune system and to define the genetic and environmental factors that affect inflammation and regulation, which could determine disease progression or nonprogression. Families that include a family member with T1D will be recruited, as well as unrelated, healthy controls as a comparison group.

Participants will have height and weight measured, complete a social & medical history questionnaire, and have blood drawn for analysis for HLA haplotype (a genetic sequence related to type 1 diabetes susceptibility)diabetes, blood glucose, immune system response, complete blood count, and autoantibody measurements. Some family members may return for follow-up visits for up to 10 years.

ELIGIBILITY:
Inclusion Criteria (Families):

* Families where at least one first-degree family member has type 1 diabetes
* The diabetic proband in the family was diagnosed before the age of 39
* Family members must be at least 2 years old to participate

Exclusion Criteria (Families):

* Families with no history of type 1 diabetes
* Families with a history of diabetes that is not type 1 (LADA, MODY, type 2 etc.)

Inclusion Criteria (Controls):

* No family history of type 1 diabetes or other autoimmune conditions
* Age 2 or older

Exclusion Criteria (Controls):

* Personal or family history of autoimmune disease

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with T1D seen at clinics at the Children's Wisconsin (n~1500) and Froedtert Hospital (n~800) will be targeted. In families with a child proband, siblings will be asked to join the study. If the diabetic child has an aunt, uncle, or cousin with T1D, then siblings in that nuclear family will also be recruited. Adult proband families will include the adult affected by T1D and their children. Adult proband families must include children <17 years of age. If the adult proband has a sibling, niece, or nephew with T1D, siblings in that nuclear family will be recruited as well. The age-of-diagnosis criterion for the proband will be less than 39 years and insulin therapy started within 5 years of diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2001-08 (Actual); Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Onset of Type 1 diabetes | Up to 10 years
  The primary outcome is the development of diabetes as defined by the American Diabetes Association (ADA) based on the presence of symptoms and unequivocal hyperglycemia.
Autoantibody Measurement | Up to 10 years
  Presence or absence of the autoantibodies related to type 1 diabetes: IA-2 (islet antigen), GAD65 (pancreatic islet cell autoantibody), IAA (insulin autoantibody), ZnT8 (zinc transporter 8)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hessner, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified samples and data will be shared with other researchers.